CLINICAL TRIAL: NCT04583774
Title: Developing a Computational Electroencephalogram (EEG) Paradigm to Study Prediction Error in Anorexia Nervosa
Brief Title: Developing an EEG Paradigm to Study Prediction Error in Anorexia Nervosa
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Guido Frank, Professor, University of California, San Diego
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 191785
Record Dates: First submitted 2020-09-25; First posted 2020-10-12 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anorexia Nervosa Group (Other): Participants with anorexia nervosa
  Interventions: Other: Prediction error tasks
- Healthy Control Group (Other): Participants who are considered to be healthy controls
  Interventions: Other: Prediction error tasks

INTERVENTIONS:
Other: Prediction error tasks — The intervention involves two tasks, one that involves taste stimuli and another that involves monetary stimuli, and test their impact o brain response in electro encephalography (EEG) and functional magnetic resonance imaging (fMRI)

SUMMARY:
Adolescent anorexia nervosa (AN) is an eating disorder associated with intense fear of weight gain, food refusal, and severe weight loss. AN is the third most common chronic illness among adolescent females with a mortality rate 12 times higher than expected for females 15-24 years old. Little is known about biomarkers in adolescent AN.

Neuroimaging studies have repeatedly suggested altered reward processing in AN including in studies using the dopamine associated prediction error (PE) model. The brain PE response is elicited during unexpected receipt or omission of reward stimuli and thought to reflect the functionality of brain dopamine circuits. This is an important research direction as the dopamine system can be manipulated pharmacologically. In ill and recovered adult AN, unexpected or randomly applied sucrose taste stimuli evoked higher insular and striatal responses and unexpected omission or receipt of monetary or taste reward was associated with a similar response pattern in adolescent AN. PE was also inversely related to weight gain in treatment. Thus, PE brain response promises to be an important biological marker for adolescent AN with predictive value for treatment outcome. However, functional brain imaging is costly, prohibitive for instance for individuals with braces or other metal in their body and only available at certain centers. In order to study PE in AN in larger scale studies, a more practical approach and method need to be developed. In this application, we will use the exploratory/developmental R21 mechanism to develop a study protocol using electroencephalography (EEG) to study PE signals in adolescent AN. Recent studies in healthy individuals support that this is a valid approach.

Our primary goal for this study is to test the feasibility of the use of EEG for prediction error and reversal learning studies in AN with the longer term goal of replacing fMRI that is costly and associated with frequent participant rule out.

In Aim 1. we test the feasibility of adapting a computational taste PE reinforcement learning paradigm from fMRI to EEG in adolescents with AN and healthy controls. We expect that we will find internal consistency of taste PE brain response across fMRI and EEG in adolescents with AN as well as age-matched healthy controls, within each group. We further expect that we will find preliminary evidence that the EEG paradigm will be able to discriminate the AN group from the HC adolescents based on feedback related negativity and higher event-related potential amplitudes, which will correlate with fMRI PE brain response.

In Aim 2., we test whether a monetary PE paradigm will show similar EEG brain response as taste PE in Aim 1. to establish the generalizability of EEG taste and non-taste paradigms.

The development of an EEG based reward PE study paradigm will enable us in the future to conduct large-scale studies that will be less costly and independent from brain imaging centers that are only available to a small subset of adolescents with AN.

ELIGIBILITY:
Inclusion Criteria:

Healthy Controls

* Females ages 11 - 17 years
* Healthy body weight between 90 and 110 % average body weight.
* Edinburgh Handedness Inventory Revised (EHI-R) LQ* score > +200
* English is primary language spoken

Restricting Type Anorexia Nervosa

* Females ages 11 - 17 years
* Diagnostic criteria. Current diagnosis of AN, including being underweight below 17.5 body mass index (BMI, kg/m2), will have a severe fear of weight gain, body image distortion and absence of the menstrual cycle over three consecutive months (if applicable).
* First 1-2 weeks in treatment at The University of California San Diego Eating Disorders Center for Treatment and Research or Rady Children's Hospital San Diego Medical Behavioral Unit.
* Restricting subtype, that is without binge/purge behaviors
* Edinburgh Handedness Inventory Revised (EHI-R) LQ* score > +200
* English is primary language spoken

Exclusion Criteria:

Healthy Controls

* Current pregnancy or breast feeding within last 3 months
* Illiterate/Blind individuals
* First degree relative with current or past eating disorder
* Current Medications other than BCP or IUD
* Past or present Axis I psychiatric disorder including substance or alcohol use disorder as determined through PI interview and MINI-Kid clinical interview
* Major Medical illness (as determined through medical history in bioscreen and PI interview) such as:

  * Conditions that are life threatening:

    * cancer
    * heart disease
    * stroke
    * HIV/AIDS
    * Seizure Disorders
  * Conditions that are life threatening Conditions that cause serious disability without necessarily being life threatening:

    * stroke
    * closed head or spinal cord injuries
    * mental retardation
    * congenital malformations.
  * Conditions that cause significant pain or discomfort that can cause serious interruptions to life activities:

    * severe allergies
    * migraine
    * arthritis
    * sickle cell disease
  * Conditions that require major commitments of time and effort from care-givers for a substantial period of time:

    * mobility disorders
    * blindness
    * Alzheimer's disease and other dementias
    * chronic obstructive pulmonary disease
    * paraplegia or quadriplegia
    * Down's syndrome
    * depression
  * Conditions that may require frequent monitoring:

    * diabetes
    * conditions requiring anticoagulation treatment
    * severe asthma
    * severe allergies
    * schizophrenia and other psychotic illnesses.
  * Conditions that predict or are associated with severe consequences:

    * hypertension (associated with heart disease)
    * depression (associated with suicide)
    * diabetes (associated with blindness, kidney failure)
    * alcohol and other substance abuse (associated with intentional and unintentional injuries).
* Recent history of suspected substance abuse or a lifetime history of psychostimulant abuse and/or dependence
* Metal implants or braces (as determined through fMRI screening form)

Anorexia Nervosa

* Pregnancy or breast feeding within last 3 months
* Lifetime history of bipolar disorder or psychosis
* Illiterate/Blind individuals
* Use of an anti-psychotic or other dopamine acting medication including stimulants within the past week at time of MRI
* Recent history of substance abuse or dependence (within the last month)
* Major Medical illness (as determined through medical history in bioscreen and PI interview) such as:

  * Conditions that are life threatening:

    * cancer
    * heart disease
    * stroke
    * HIV/AIDS
    * Seizure Disorders
  * Conditions that are life threatening Conditions that cause serious disability without necessarily being life threatening:

    * stroke
    * closed head or spinal cord injuries
    * mental retardation
    * congenital malformations.
  * Conditions that cause significant pain or discomfort that can cause serious interruptions to life activities:

    * severe allergies
    * migraine
    * arthritis
    * sickle cell disease
  * Conditions that require major commitments of time and effort from care-givers for a substantial period of time:

    * mobility disorders
    * blindness
    * Alzheimer's disease and other dementias
    * chronic obstructive pulmonary disease
    * paraplegia or quadriplegia
    * Down's syndrome
  * Conditions that may require frequent monitoring:

    * diabetes
    * conditions requiring anticoagulation treatment
    * severe asthma
    * severe allergies
    * schizophrenia and other psychotic illnesses.
  * Conditions that predict or are associated with severe consequences:

    * hypertension (associated with heart disease)
    * diabetes (associated with blindness, kidney failure)
    * alcohol and other substance abuse (associated with intentional and unintentional injuries) within the last month
* Metal implants or braces (as determined through fMRI screening form)

Ages: 11 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Correlation between Reward Prediction Error Brain Response using functional Magnetic Resonance Imaging (fMRI) and Electroencephalography (EEG) | Immediate during brain scanning
  Study participants will undergo an fMRI session during which they perform a taste reward prediction error paradigm. Blood oxygen-level dependent (BOLD) functional activity will be acquired during the task. The prediction error signal will be modeled based on trial sequence. The same individuals will perform the prediction error task during EEG. fMRI and EEG results for brain regions will be compared and tested for correlations between modalities.
Reward Prediction Error Brain Response using Electroencephalography (EEG) to separate healthy controls from individuals with anorexia nervosa. | Immediate during brain scanning
  We will test whether regional brain EEG recordings from the taste prediction error paradigm in Outcome 1 can distinguish individuals with anorexia nervosa from healthy controls.
Monetary Reward Prediction Error Brain Response using EEG will show similar regional brain response compared to taste prediction error response. | Immediate during brain scanning
  Study participants will undergo an EEG session during which they perform a monetary reward prediction error paradigm. The results will be compared to the taste paradigm results from Outcome 1.

CONTACTS AND LOCATIONS:
Overall Officials: Guido Frank, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

DOCUMENTS (1):
  • Informed Consent Form (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/74/NCT04583774/ICF_000.pdf